CLINICAL TRIAL: NCT02864862
Title: Esthetic Outcomes Following Immediate Implant Combine With Soft Tissue Augmentation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Chun-Teh Lee, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-DB-16-0286
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Results first posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-11

CONDITIONS: Dental Implant; Immediate Dental Implant; Soft Tissue Augmentation
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Immediate implant (Active Comparator): Immediate implant alone
  Interventions: Device: Immediate implant
- Immediate implant combined with SCTG (Active Comparator): Subepithelial connective tissue graft (SCTG)
  Interventions: Device: Immediate implant; Biological: SCTG
- Immediate implant combined with ADM (Active Comparator): Acellular dermal matrix (ADM)
  Interventions: Device: Immediate implant; Biological: ADM

INTERVENTIONS:
Device: Immediate implant
Biological: SCTG
  Arms: Immediate implant combined with SCTG
Biological: ADM
  Arms: Immediate implant combined with ADM

SUMMARY:
The purpose of this study is to evaluate the esthetic outcomes following immediate implant combined with the autogenous tissue graft or acellular dermal matrix compared to immediate implant alone.

ELIGIBILITY:
Inclusion Criteria:

* patients who are in need of a tooth extraction at the maxillary premolar, canine and incisor region, and subsequent single implant placement.
* The reasons for extraction will include poor endodontic prognosis and/or unrestorable teeth (extensive caries, traumatic fractures, fractures of endodontically treated teeth, root perforation, root resorption with or without radiographic periapical lesion up to 3 mm in diameter). patients who are systemically healthy or with controlled common systemic conditions (controlled hypertension, controlled diabetes HbA1c up to 7 %).
* adjacent teeth have to be present and the eligible tooth has esthetically acceptable buccal gingival margin position prior to surgery, compared to neighboring teeth and contralateral tooth, and adequate width of buccal keratinized gingiva(≥3mm).
* level of radiographic bone level has the distance from CEJ to interproximal crest up to 4 mm.
* Location of buccal alveolar crest has to be generally within 4 mm from the free gingival margin, verified after the extraction, before randomization; and fenestration, if present, up to 3mm in diameter at the apical part of the root and affecting less than 30% of the buccal socket wall.

Exclusion Criteria:

* currently smoke exceeding 10 cigarettes/ day
* severe parafunctional habits, malocclusion or intent of orthodontic therapy in the future and are pregnant.
* teeth in the surgical site will be excluded if there is advanced periodontal disease or periapical lesion causing significant bony defects that are beyond the criteria mentioned at Section 3.3.
* allergy to antibiotics contained in the ADM (Gentimicin, Cefoxitin, Lincomcin, polymixin B and Vancomycin) will not be included in the immediate implant combined with ADM group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Teh Lee, DDS, DMSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Jung M, Tran D, Chang CC, Kim SK, Tsukiboshi Y, Min S, Ayilavarapu S, Lee CT. Volumetric buccal bone alterations at immediate implant sites with or without soft tissue augmentation: A 6-month assessment. J Periodontol. 2025 Aug 10. doi: 10.1002/jper.11381. Online ahead of print. PMID 40785129

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Implant Combined With SCTG: Immediate implant plus Subepithelial connective tissue graft (SCTG)
- Immediate Implant Combined With ADM: Immediate implant plus Acellular dermal matrix (ADM)
Period: Overall Study
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Started | 15 | 15 | 16
Received Intervention | 15 | 15 | 16
3-month Follow up | 15 | 15 | 16
6-month Follow up | 15 | 15 | 15
12-month Follow up | 14 | 15 | 14
Completed | 14 | 15 | 14
Not Completed | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant | Total
Number analyzed (Participants) | 15 | 15 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.53 (9.81) | 63.53 (13.16) | 58.88 (11.55) | 61.26 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 9 | 24
  Male | 8 | 7 | 7 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 16 | 46
Number of participants that smoke [Count of Participants; unit: Participants] | 1 | 0 | 4 | 5
Number of participants that have diabetes [Count of Participants; unit: Participants] | 6 | 2 | 0 | 8
Number of participants that have hypertension [Count of Participants; unit: Participants] | 3 | 5 | 5 | 13
Number of participants with anterior implant sites [Count of Participants; unit: Participants] | 7 | 6 | 9 | 22
Number of participants with pre molar implant sites [Count of Participants; unit: Participants] | 8 | 9 | 7 | 24
Implant diameter [Count of Participants; unit: Participants]
  3.5 millimeters (mm) | 6 | 4 | 7 | 17
  4.3mm | 8 | 11 | 9 | 28
  5.0mm | 1 | 0 | 0 | 1
Implant length [Count of Participants; unit: Participants]
  10mm | 0 | 3 | 0 | 3
  11.5mm | 4 | 7 | 4 | 15
  13mm | 8 | 5 | 8 | 21
  16mm | 3 | 0 | 4 | 7
Mean probing depth(PD) of the tooth [Mean (Standard Deviation); unit: millimeters] | 2.28 (0.47) | 2.29 (0.38) | 2.24 (0.45) | 2.26 (0.43)
Mean number of sites on tooth with bleeding on probing (BOP) [Mean (Standard Deviation); unit: number of sites] | 2.47 (1.68) | 2.60 (1.72) | 2.44 (1.59) | 2.50 (1.66)
Mean number of sites on tooth with plaque (PL) [Mean (Standard Deviation); unit: number of sites] | 4.20 (1.66) | 4.13 (2.13) | 4.63 (1.54) | 4.32 (1.78)
Width of keratinized tissue at baseline [Mean (Standard Deviation); unit: millimeters] | 4.70 (1.16) | 4.83 (1.32) | 4.50 (1.20) | 4.67 (1.22)
Preoperative buccal soft tissue thickness [Mean (Standard Deviation); unit: millimeters] | 1.24 (0.25) | 1.34 (0.25) | 1.18 (0.31) | 1.25 (0.27)
Postoperative buccal soft tissue thickness [Mean (Standard Deviation); unit: millimeters] | 2.38 (0.32) | 2.57 (0.30) | 1.18 (0.31) | 2.02 (0.31)
Peri-implant marginal bone level [Mean (Standard Deviation); unit: millimeters]
  Mesial | -0.11 (0.31) | -0.08 (0.31) | -0.31 (0.83) | -0.169 (0.55)
  Distal | -0.03 (0.10) | -0.95 (2.30) | -0.36 (1.21) | -0.44 (1.49)
Peri-implant crestal bone level [Mean (Standard Deviation); unit: millimeters]
  Mesial | 3.59 (1.09) | 3.01 (1.08) | 3.56 (1.27) | 3.39 (1.15)
  Distal | 3.02 (1.21) | 2.88 (1.13) | 3.31 (1.19) | 3.07 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Change in Ridge Dimension
Description: Change in ridge dimension is calculated as the value at 6 months minus the value at baseline. To take ridge dimension measurements, impressions were taken at baseline and 6 months, models were made from these impressions, the models were scanned, and then ridge dimension of scanned models was assessed using software. Ridge dimension was assessed at (and at 1mm increments below) the initial soft tissue margin.
Time Frame: baseline, 6 months after surgery
Population: Data were not collected for one participant in the immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 15 | 15 | 15
millimeters (mm)
  Initial soft tissue margin | -1.65 (1.27) | -1.87 (1.19) | -1.44 (0.98)
  1mm below initial soft tissue margin | -1.37 (0.79) | -1.60 (0.93) | -1.41 (0.64)
  2mm below initial soft tissue margin | -0.87 (0.71) | -1.01 (0.66) | -1.23 (0.61)
  3mm below initial soft tissue margin | -0.47 (0.62) | -0.65 (0.66) | -1.06 (0.66)
  4mm below initial soft tissue margin | -0.15 (0.51) | -0.37 (0.74) | -0.86 (0.63)
  5mm below initial soft tissue margin | 0.14 (0.61) | -0.17 (0.84) | -0.64 (0.65)

2. Primary Outcome: Change in Ridge Dimension
Description: Change in ridge dimension is calculated as the value at 12 months minus the value at baseline. To take ridge dimension measurements, impressions were taken at baseline and 12 months, models were made from these impressions, the models were scanned, and then ridge dimension of scanned models was assessed using software. Ridge dimension was assessed at (and at 1mm increments below) the initial soft tissue margin.
Time Frame: baseline, 12 months after surgery
Population: Data were not collected for 1 participant in the Immediate implant combined with SCTG arm and 2 participants in the Immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 14 | 15 | 14
millimeters (mm)
  Initial soft tissue margin | -1.80 (1.52) | -2.33 (1.15) | -1.91 (0.94)
  1mm below initial soft tissue margin | -1.21 (0.92) | -1.61 (0.95) | -1.54 (0.81)
  2mm below initial soft tissue margin | -0.87 (0.75) | -1.08 (0.66) | -1.27 (0.75)
  3mm below initial soft tissue margin | -0.48 (0.63) | -0.78 (0.65) | -1.21 (0.82)
  4mm below initial soft tissue margin | -0.23 (0.60) | -0.51 (0.55) | -1.11 (0.85)
  5mm below initial soft tissue margin | -0.02 (0.61) | -0.41 (0.55) | -0.90 (0.79)

3. Secondary Outcome: Change in Gingival Level
Description: Change in gingival level is calculated as the value at 6 months minus the value at baseline. Gingival level is measured at three sites: mesial, mid-buccal and distal sites. Gingival level is measured from a notch on a custom fabricated stent to the mucosal margin.
Time Frame: baseline, 6 months after surgery
Population: Data were not collected for one participant in the immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 15 | 15 | 15
millimeters (mm)
  Mesial | -0.47 (0.61) | -0.9 (1.24) | -0.67 (0.70)
  Mid-buccal | 0.2 (0.90) | -0.37 (1.03) | 0.3 (0.94)
  Distal | -0.23 (0.62) | -0.70 (0.92) | -0.43 (0.94)

4. Secondary Outcome: Change in Gingival Thickness
Description: Change in gingival thickness is calculated as the value at 6 months minus the value at baseline. Gingival thickness is measured using a stoppered endodontic file (#30) penetrating through the facial soft tissue 3 millimeters (mm) below the mid-buccal peri-implant mucosal margin.
Time Frame: baseline, 6 months after surgery
Population: Data were not collected for one participant in the immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 15 | 15 | 15
millimeters (mm) | 0.86 (0.25) | 0.97 (0.47) | 0.14 (0.14)

5. Secondary Outcome: Change in Width of Keratinized Gingiva
Description: Change in width of keratinized gingiva is calculated as the value at 6 months minus the value at baseline.
Time Frame: baseline, 6 months after surgery
Population: Data were not collected for one participant in the immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 15 | 15 | 15
millimeters (mm) | 0.27 (0.73) | -0.47 (1.06) | 0.37 (0.85)

6. Secondary Outcome: Change in Alveolar Bone Level (Marginal)
Description: Change in alveolar bone level is calculated as the value at 6 months minus the value at baseline. The bone level measurement, taken from the standardized periapical radiographs, was defined as the distance from the first bone to implant contact (IB) at either the mesial or the distal aspect of the implant to the implant platform. Specifically, marginal bone level was defined as the distance between the vertical implant bone level (IB; the first bone to implant contact) and implant platform (IP). Crestal bone level was defined as the distance between the interproximal crestal bone level (IC) and implant platform (IP).
Time Frame: baseline, 6 months after surgery
Population: Data were not collected for one participant in the immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 15 | 15 | 15
millimeters (mm)
  Mesial | -0.45 (0.78) | -0.70 (0.90) | -0.37 (1.05)
  Distal | -0.19 (0.62) | -0.27 (2.63) | -0.40 (1.69)

7. Secondary Outcome: Change in Alveolar Bone Level (Crestal)
Description: Change in alveolar bone level is calculated as the value at 6 months minus the value at baseline. The bone level measurement, taken from the standardized periapical radiographs, was defined as the distance from the first bone to implant contact (IB) at either the mesial or the distal aspect of the implant to the implant platform. Specifically, crestal bone level was defined as the distance between the interproximal crestal bone level (IC) and implant platform (IP).
Time Frame: baseline, 6 months after surgery
Population: Data were not collected for one participant in the immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 15 | 15 | 15
millimeters (mm)
  Mesial | -0.62 (1.64) | -0.35 (0.81) | -0.43 (0.95)
  Distal | -0.88 (1.22) | -0.74 (1.10) | -0.78 (0.87)

8. Secondary Outcome: Change in Bone Dimension
Description: Change in bone dimension is calculated as the value at 6 months minus the value at baseline. To measure bone dimensions, bone dimensions on cone beam computed tomography (CBCT) images were assessed using software. Bone dimension was assessed at the initial buccal crestal bone level (and at 1mm increments below).
Time Frame: baseline, 6 months after surgery
Population: Data were not collected for one participant in the immediate implant arm.
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
Number analyzed (Participants) | 15 | 15 | 15
millimeters (mm)
  Initial buccal crestal bone level | -1.34 (1.03) | -0.85 (0.92) | -0.77 (0.79)
  1mm below initial crestal bone level | -1.74 (0.94) | -1.40 (1.39) | -1.33 (1.11)
  2mm below initial crestal bone level | -1.40 (0.92) | -0.93 (1.20) | -1.10 (0.82)
  3mm below initial crestal bone level | -0.86 (0.47) | -0.79 (1.10) | -0.67 (0.56)
  4mm below initial crestal bone level | -0.76 (0.43) | -0.71 (0.93) | -0.48 (0.50)
  5mm below initial crestal bone level | -0.62 (0.48) | -0.66 (0.69) | -0.46 (0.47)
  6mm below initial crestal bone level | -0.56 (0.52) | -0.75 (0.57) | -0.58 (0.51)
  7mm below initial crestal bone level | -0.44 (0.56) | -0.59 (0.45) | -0.56 (0.46)
  8mm below initial crestal bone level | -0.52 (0.56) | -0.50 (0.30) | -0.58 (0.51)
  9mm below initial crestal bone level | -0.46 (0.54) | -0.28 (0.34) | -0.47 (0.48)
  Coronal third | -1.34 (0.65) | -0.99 (0.98) | -0.97 (0.63)
  Middle third | -0.65 (0.43) | -0.71 (0.69) | -0.51 (0.48)
  Apical third | -0.47 (0.53) | -0.46 (0.32) | -0.54 (0.45)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Immediate Implant Combined With SCTG | Immediate Implant Combined With ADM | Immediate Implant
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT02864862/Prot_SAP_000.pdf